CLINICAL TRIAL: NCT04645134
Title: Physical Activity and Cognitive Function in Older Adults: A Novel Role for GPLD1
Acronym: BrainFit
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Eric Ravussin, Associate Executive Director for Clinical Science, Pennington Biomedical Research Center
Other Study IDs: PBRC 2020-050
Record Dates: First submitted 2020-11-22; First posted 2020-11-27 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Aging; Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inactive: Older adults who have a sedentary or under-active lifestyle.
  Interventions: Behavioral: Brain Health Assessments
- Highly Active: Older adults who have a highly active lifestyle.
  Interventions: Behavioral: Brain Health Assessments

INTERVENTIONS:
Behavioral: Brain Health Assessments — The investigators are enrolling up to 28 healthy, older adults (ages 65-85 y, BMI 20-35 kg/m2) stratified by current physical activity level (equal inactive vs. equal highly active). Each physical activity group (inactive and highly active) will undergo a blood draw, body composition, resting metabolic rate, cognitive testing, and magnetic resonance (MR) imaging.

SUMMARY:
The investigators are conducting a cross-sectional, observational study to investigate whether plasma GPLD1 concentrations are associated with higher cognitive function and better brain structure and function in two groups of older adults with high or low levels of physical activity.

DETAILED DESCRIPTION:
This is a cross-sectional, observational study which will enroll up to 28 healthy, older adults (65-85 y, BMI 20-35 kg/m2), and stratify by current self-reported physical activity level (equal inactive vs. equal highly active).

Aim 1: Investigate whether physical activity level is associated with GPLD1.

Aim 2: Investigate whether cognitive function and brain structure/function are associated with GPLD1.

ELIGIBILITY:
Inclusion Criteria:

* Ages 65-85 y (inclusive)
* Body mass index (BMI) of 20-35 kg/m2 (inclusive)
* Willing to have blood and data stored for future research use

Exclusion Criteria:

* History of clinically diagnosed diabetes (Type 1 or 2) or a fasting blood glucose >126 mg/dL
* Diagnosed Alzheimer's disease, dementia, or related-brain diseases
* Chronic use of atypical antipsychotic or bipolar medications
* Initiation of novel pharmacotherapy agents (such as antidepressant, hypertension, or dyslipidemia) within the last 3 months
* Uncontrolled hypertension (blood pressure >160 systolic or >110 diastolic)
* Asthma that limits the ability to participate in moderate to vigorous physical activity or requiring systemic glucocorticoid administration
* Emphysema that limits the ability to participate in moderate to vigorous physical activity or requiring systemic glucocorticoid administration
* Current alcohol use exceeding 14 drinks per week in women, exceeding 21 drinks per week in men, having treatment for alcohol abuse in the last year, or having treatment for alcohol abuse more than 1 year ago (but with inability to refrain from alcohol in the past year)
* Use of illegal drugs or marijuana within 1-month of completing a Screening Visit; treatment for drug addiction in the 1-year or having treatment for drug addiction >1-year ago, but with an inability to refrain from the drug of addiction in the 1-year
* Unwilling to abstain from illegal drugs and marijuana for the duration of the study
* Contraindication for MRI (e.g., metal objects, claustrophobia, etc.)
* Psychotic mental illness (e.g., schizophrenia, bipolar, on-and- off use of anti-psychotic medication)
* History of cardiovascular disease (or diseases of the heart, lungs, or blood) that limits participation in moderate to vigorous physical activity
* History of liver, blood, kidney, thyroid or other diseases that limits moderate to vigorous physical activity at the time of enrollment
* Cancer that limits moderate to vigorous physical activity
* Treatment with systemic immunosuppressant medication
* Taking adrenergic stimulants (e.g., amphetamine) or adrenergic blockers (e.g., Propanolol) that will alter metabolic rate
* Have plans to substantially alter their current level of physical activity over the next 1-month

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Up to 28 healthy, older adults (ages 65-85 y, BMI 20-35 kg/m2) stratified by current physical activity level will be enrolled. The investigators will enroll an equal number of inactive adults and an equal number of highly active adults.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of GPLD1 | 1 day
  Plasma GPLD1 (by a blood draw) is performed.

SECONDARY OUTCOMES:
Physical activity level | 7 days
  Physical activity level assessment (by accelerometry) is performed.
Total grey matter volume | 1 day
  Total grey matter volume (by structural MRI) is performed.
Brain activity and function | 1 day
  Brain activity and function (by functional MRI) during execution of two cognitive tasks (Stroop Task and Attention Network Task (ANT)) is performed.
Cognitive function | 1 day
  Cognitive function testing (using the NIH Toolbox Cognitive Battery) is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Marlatt, PhD, MPH, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Marlatt KL, Lowe AC, Sanchez-Delgado G, Beyl RA, Viverito MK, Keller JN, Carmichael OT, Ravussin E. Associations between physical activity, brain health, cognitive function, and circulating GPLD1 in healthy older (65-85 years) individuals. Geroscience. 2025 Jun;47(3):3821-3834. doi: 10.1007/s11357-024-01459-8. Epub 2025 Jan 6. PMID 39762691